CLINICAL TRIAL: NCT03078868
Title: Utility of Diffusion-weighted MR Imaging in Guiding Selective Percutaneous Drainage of Postoperative Intra-abdominal Abscesses After Colorectal Resection
Brief Title: Utility of Diffusion-weighted MR Imaging
Acronym: DWMRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of accrual and PI left institution
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB16-1771
Record Dates: First submitted 2017-02-23; First posted 2017-03-14 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: DWM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single-point intervention (Experimental): magnetic resonance scanner
  Interventions: Device: Magnetic Resonance Scanner

INTERVENTIONS:
Device: Magnetic Resonance Scanner — MRI

SUMMARY:
To determine whether DW-MRI is applicable in the evaluation of post-operative collections, and whether utilization of DW-MRI can enhance application of percutaneous drainage and prevent unnecessary drainage.

DETAILED DESCRIPTION:
Percutaneous drainage of intra-abdominal abscesses occurring as a complication of colon and rectal resection has been a major advance in the management of surgical patients. Proper patient selection is critical for safe and effective management in this population. Almost ¾ of patients undergoing CT scan after colorectal resection due to clinical suspicion of intrabdominal process will have at least one fluid collection identified. These collections can represent a spectrum of clinical entities and there is not a consensus on the most effective management of these collections or even the definition of abscess. Currently, reliance on radiologic criteria in isolation can lead to overuse of interventional procedures. For example, 40% of rim-enhancing collections are sterile on aspiration. The surgeons' clinical suspicion for abscess and radiologic proximity to an anastomosis are the only criteria that are useful in predicting abscess versus sterile collection. A further consideration is the natural history of these abscesses. Studies in the diverticulitis literature have demonstrated that abscesses less than 3 cm in greatest dimension are successfully managed with antibiotics alone, while abscesses greater than 6.5 cm are likely to require intervention. However, this leaves a great number of abscesses between 3 cm and 6.5 cm that fall into uncertain grounds. In contrast to diverticulitis, where it can be reasonably inferred that an associated abdominopelvic collection is indeed and abscess, management of fluid collections identified post-operatively and determination of who will benefit from drainage is less clear. A novel radiologic technique with high discrimination between sterile and infected collection would be of great clinical utility in the post-operative management of fluid collections after colorectal resection.

The proposed research project seeks to broaden applicability of a proven but rarely used method, diffusion weighted magnetic resonance imaging (DW-MRI), to discriminate sterile or benign from infected abdominopelvic fluid collections, in order to enhance the utilization of percutaneous drainage in the post-operative setting after colorectal resection. Ability to streamline a limited MRI protocol to efficiently obtain diffusion weighted imaging of the abdominal cavity will be key to applying this methodology into daily practice. Secondly, it is not known whether DW-MRI can effectively discriminate specifically post-operative sterile collections from abscesses. This is one of the primary aims of this pilot study and will be used to generate hypothesis for a full-scale study.

Adult patients who have undergone a colon or rectal resection at the University of Chicago Medicine and have developed a CT-proven abdominopelvic fluid collection > 3 cm in greatest dimension will be eligible for inclusion in the study. The surgeon will then determine using traditional clinical and radiologic factors whether percutaneous drainage is desired. All patients with discrete abdominopelvic fluid collections > 3 cm in greatest dimension will undergo DW-MRI, and then be taken directly to the interventional radiology suite for drainage, or continue best medical care if drainage is felt to be unnecessary. Fluid will be sent for culture and gram stain, as well as cell count. In addition, the interventional radiology team will qualify the fluid in their notation as 'purulent', 'serous', 'sanguinous', etc.. Any patients initially managed without drainage who fail this medical management and ultimately undergo percutaneous drainage will be considered the crossover group.

DW-MRI readings will be analyzed and ADC values will be compared and validated in an attempt to report a threshold apparent diffusion coefficient (ADC) that reliably discriminates sterile and infected post-operative fluid collections. The effect size from utilization of DW-MRI (defined as a change in management decision to pursue drainage or hold on drainage) to determine if this is a useful clinical tool. Because it is not yet know how DW-MRI should be interpreted in this clinical setting, the DW-MRI acquisition will not be utilized in any way in the clinical care of the study patients. The DW-MRI data is considered a single-point intervention and will only be used to define an ADC threshold that can discriminate sterile from infected collections. The data will help us to identify potential limitations of DWI in differentiation of abscess from non-infected collections and allow us to determine the appropriate cohort size for a future clinical trial. Based on the correlation with DWI and clinical data, we will explore and suggest novel acquisition and analysis methods for quantitative DWI.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients who have undergone a colon or rectal resection at UCM and have developed a CT-proven abdominopelvic fluid collection > 3 cm in greatest dimension

Exclusion Criteria:

• Adult patients who have not undergone a colon or rectal resection at UCM and have developed a CT-proven abdominopelvic fluid collection > 3 cm in greatest dimension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Cannon, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
N/A-data won't be shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single-point Intervention
Started | 3
Completed | 0
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: Study terminated for lack of accrual and PI left institution
Arm/Group | Single-point Intervention
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender information was not collected Population: Gender information/data not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Apparent Diffusion Coefficient (ADC) From Infected Post-operative Fluid Collections
Description: Two radiologists will independently review the MR images for detection of collections. ADC maps will be generated for each patient. Each radiologist will assign a 1-5 point score based on the level of confidence in the diagnosis of abscess. These radiologists will then measure ADC of the collections in each patient on ADC maps. Mean and 10th percentile ADC values will be computed by placement of region of interest (ROI) on ADC maps using DW images as guide. Each ROI will be placed in the center of the collection over the darkest pixels on ADC maps keeping size as large as possible and avoiding the volume averaging from the surrounding tissue. The reference standard for the diagnosis of abscess will be based on the analysis of aspiration fluid from the collection. Following statistical analysis, an ROC curve will be constructed for ADC values, and area under the curve measured forthe overall ability of ADC in differentiation of abscess from non-infected collections
Time Frame: 1 year
Population: study terminated for lack of accrual and PI left institution
Arm/Group | Single-point Intervention
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: not collected - study terminated for lack of accrual and PI left institution
Description: not data collected - study terminated for lack of accrual and PI left institution
Arm/Group | Single-point Intervention
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This trial was terminated for lack of accrual, so no data was collected and the Principal Investigator left the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT03078868/Prot_SAP_000.pdf